Appendix 1: Template of clinical research plan

Project source and number: Self-selected topic

## Plastic surgery clinical research project

Leader Unit: Xijing Hospital

Project Leader: Xianjie Ma

**Department:**Plastic surgery

Tel:+86 29 8477 5301

E-mail:majing@fmmu.edu.cn

Participating Unit: Xijing Hospital

Study Period: Jan 01,2018-Jan 01,2020

Version Number: V 2.0

Version date:Dec 08,2017

## **Summary project**

## - Research Program

| Project name | Comparison of clinical efficacy of golden microneedles and |
|---|---|
| | 1565nm non-ablative dot matrix laser in the treatment of eyelid |
| | pouches |
| Purpose of the | The purpose of this test is to compare the efficacy of golden |
| Study | microneedles and 1565nm non-ablative dot matrix laser in the |
| Study | treatment of eyelid pouches. |
| Type of study | Randomized, double-blind, self-controlled study |
| Number of cases | 16 |
| | Inclusion Criteria: |
| | 1. Patients with blepharoplasty; |
| | 2. Fitzpatrick III-V; |
| | 3. Males and females between 18-60 years old. |
| | Exclusion criteria: |
| Inclusion and | 1. Other diseases that can cause pathological changes in |
| | periorbital soft tissue, such as collagen disease, kidney disease, |
| | liver cirrhosis, Graves disease, diabetes, scleroderma, |
| Exclusion | hyperlipidemia, myasthenia gravis, Horner syndrome, |
| Criteria | myosermatitis etc; |
| | 2. Other diseases affecting wound healing, such as systemic |
| | diseases such as diabetes, heart disease, hypertension, infectious |
| | diseases such as tuberculosis, hepatitis, skin diseases, tumors, |
| | etc.; such as dry eye syndrome, cataract, glaucoma ophthalmic |
| | diseases. |
| | 3. Take steroids, vasodilators, anticoagulants (warfarin, non- |
| | steroidal anti-inflammatory drugs, aspirin, heparin, etc.) and |
| | retinoids 2 weeks before surgery. Local infections on the skin. |

| | 4.Patients with blepharoplasty, periorbital laser, botulinum toxin |
|---|---|
| | type A treatment history, and herpes simplex virus (HSV) |
| | infection history 6 months before surgery. History of exposure 2 |
| | months before surgery. |
| | 5.Scar physical, pregnancy, bilateral asymmetrical eye bags. |
| | Before entering the group, they were informed of their risks, |
| | benefits, and possible complications after the operation, and |
| | signed an informed consent. |
| | 6.Can not guarantee treatment on time, those who fail to |
| | cooperate. |
| | 16 patients with blepharoplasty bags, and two bilateral |
| | blepharoplasty bags were treated with laser respectively, and |
| | subjective adverse reactions (pain, burning, and burnout) were |
| Treatment | recorded before treatment, 4 weeks after each treatment, and 12 |
| options | and 24 weeks after the third treatment. Itching, dryness), |
| | objective adverse reactions (erythema, pimples, edema, |
| | exudation, bleeding, scabbing, infection), patient satisfaction |
| | VAS score, visa skin tester, 3D skin test, ultrasound |
| | measurement of lower eyelid fat volume every 4 weeks Treat |
| | once and treat three times per person. |
| | Effectiveness evaluation indicators: |
| | 1.Patient satisfaction |
| | 2.Wrinkles, texture and pores by VISIA |
| Efficacy | 3.3D data changes |
| evaluation | 4.Ultrasound measurement of BLEs volume. |
| | Safety evaluation indicators: |
| | 1. Subjective adverse reactions-pain, burning, itching, dryness |
| | 2.Objective adverse reactions-erythema, pimples, edema, |
| | exudation, bleeding, crusting, infection. |
| Statistical | The pain of the left and right lower eyelids was tested by paired t |

| | methods | test, the changes of various indexes of visia, 3D, and ultrasound |
|---|---|---|
| | | were compared with the Wilcoxon symbol rank test of paired |
| | | samples, and the subjective and objective adverse reactions were |
| | | tested by $\chi^2$ test. |
| - | Study period | 2 years |

## 二、Research process

